CLINICAL TRIAL: NCT03586869
Title: QUILT-3.080: Phase 1B/2 Trial Of The NANT Pancreatic Cancer Vaccine As Treatment For Subjects With Pancreatic Cancer Who Have Progressed on or After Standard-Of-Care Therapy
Brief Title: QUILT-3.080: NANT Pancreatic Cancer Vaccine
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study halted prematurely and will not resume; participants are no longer being examined or receiving intervention
Sponsor: ImmunityBio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QUILT-3.080
Record Dates: First submitted 2018-06-22; First posted 2018-07-16 (Actual); Results first posted 2024-08-27 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2019-07

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — ALT-803; yeast-CEA vaccine; Bevacizumab; Capecitabine; Cyclophosphamide; Fluorouracil; Leucovorin; 130-nm albumin-bound paclitaxel; Oxaliplatin; avelumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- NANT Pancreatic Cancer Vaccine (Experimental): A combination of agents were administered to subjects in this study: Aldoxorubicin HCl, ALT-803, ETBX-011 (CEA), ETBX-021 (HER2), ETBX-051 (Brachyury), ETBX-061 (MUC1), GI-4000, GI-6207, GI-6301, haNK for infusion, avelumab, bevacizumab, capecitabine, cyclophosphamide, fluorouracil, leucovorin, nab-paclitaxel, oxaliplatin, and Stereotactic Body Radiation Therapy (SBRT).
  Interventions: Drug: Aldoxorubicin HCl; Biological: ALT-803; Biological: ETBX-011; Biological: ETBX-021; Biological: ETBX-051; Biological: ETBX-061; Biological: GI-4000; Biological: GI-6207; Biological: GI-6301; Biological: haNK for infusion; Biological: bevacizumab; Drug: Capecitabine; Drug: Cyclophosphamide; Drug: Fluorouracil; Drug: Leucovorin; Drug: nab-Paclitaxel; Drug: Oxaliplatin; Biological: Avelumab; Procedure: SBRT

INTERVENTIONS:
Drug: Aldoxorubicin HCl — Aldoxorubicin Hydrochloride
Biological: ALT-803 — Recombinant human super agonist interleukin-15 (IL-15) complex
Biological: ETBX-011 — Ad5 [E1-, E2b-]-CEA
Biological: ETBX-021 — Ad5 [E1-, E2b-]-HER2
Biological: ETBX-051 — Ad5 [E1-, E2b-]-Brachyury
Biological: ETBX-061 — Ad5 [E1-, E2b-]-MUC1
Biological: GI-4000 — RAS yeast
Biological: GI-6207 — Carcinoembryonic Antigen (CEA) yeast
Biological: GI-6301 — Brachyury yeast
Biological: haNK for infusion — NK-92 [CD16.158V, ER IL-2]
Biological: bevacizumab — Recombinant human anti-Vascular Endothelial Growth Factor (VEGF) IgG1 monoclonal
Drug: Capecitabine — 5'-deoxy-5-fluoro-N-[(pentyloxy) carbonyl]-cytidine
Drug: Cyclophosphamide — 2-[bis(2-chloroethyl)amino]tetrahydro-2H-1,3,2-oxazaphosphorine 2-oxide monohydrate
Drug: Fluorouracil — 5-fluoro-2,4 (1H,3H)-pyrimidinedione
Drug: Leucovorin — L-Glutamic acid, N-[4-[[(2-amino-5-formyl-1,4,5,6,7,8-hexahydro-4-oxo-6-pteridinyl)methyl]amino]benzoyl]-, calcium salt
Drug: nab-Paclitaxel — Benzenepropanoic acid, β-(benzoylamino)-α-hydroxy-(2aR, 4S, 4aS, 6R, 9S, 11S, 12S, 12aR, 12bS)-6,12b-bis(acetyloxy)-12-(benzoyloxy)-2a, 3, 4, 4a, 5, 6, 9, 10, 11, 12, 12a, 12b-dodecahydro-4,11-dihydroxy-4a, 8, 13, 13-tetramethyl-5-oxo-7,11-methano-1H-cyclodeca[3,4]benz[1,2-b]oxet-9-y1ester,(αR,βS)-(9CI) bound to albumin
Drug: Oxaliplatin — cis-[(1 R,2 R)-1,2-cyclohexanediamine-N,N'] [oxalato(2-)- O,O'] platinum
Biological: Avelumab — Recombinant human anti-programmed death-ligand 1 (PD-L1) IgG1 monoclonal antibody
Procedure: SBRT — Stereotactic Body Radiation Therapy

SUMMARY:
This is a phase 1b/2 study to evaluate the safety and efficacy of metronomic combination therapy in subjects with pancreatic cancer who have progressed on or after previous Standard of Care (SoC) chemotherapy.

DETAILED DESCRIPTION:
Treatment will be administered in two phases, an induction and a maintenance phase, as described below. Subjects will continue induction treatment for up to 1 year. Treatment in the study will be discontinued if the subject experiences progressive disease (PD) or unacceptable toxicity (not corrected with dose reduction), withdraws consent, or if the Investigator feels it is no longer in the subject's best interest to continue treatment. Those who have a complete response (CR) in the induction phase will enter the maintenance phase of the study. Subjects who experience ongoing stable disease (SD) or an ongoing partial response (PR) at 1 year may enter the maintenance phase at the Investigator's discretion. Subjects may remain on the maintenance phase of the study for up to 1 year. Treatment will continue in the maintenance phase until the subject experiences PD or unacceptable toxicity (not corrected with dose reduction), withdraws consent, or if the Investigator feels it is no longer in the subject's best interest to continue treatment. The maximum time on study treatment, including both the induction and maintenance phases, is 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old.
2. Able to understand and provide a signed informed consent that fulfills the relevant IRB or Independent Ethics Committee (IEC) guidelines.
3. Histologically-confirmed pancreatic adenocarcinoma with progression on or after SoC therapy.
4. ECOG performance status of 0 to 2.
5. Have at least 1 measurable lesion of ≥ 1.0 cm.
6. Must have a recent formalin-fixed, paraffin-embedded (FFPE) tumor biopsy specimen following the conclusion of the most recent anticancer treatment and be willing to release the specimen for prospective and exploratory tumor molecular profiling. If an historic specimen is not available, the subject must be willing to undergo a biopsy during the screening period, if considered safe by the Investigator. If safety concerns preclude collection of a biopsy during the screening period, a tumor biopsy specimen collected prior to the conclusion of the most recent anticancer treatment may be used.
7. Must be willing to provide blood samples prior to the start of treatment on this study for prospective tumor molecular profiling and exploratory analyses.
8. Must be willing to provide a tumor biopsy specimen 8 weeks after the start of treatment for exploratory analyses, if considered safe by the Investigator.
9. Ability to attend required study visits and return for adequate follow-up, as required by this protocol.
10. Agreement to practice effective contraception for female subjects of child-bearing potential and non-sterile males. Female subjects of child-bearing potential must agree to use effective contraception for up to 1 year after completion of therapy, and non- sterile male subjects must agree to use a condom for up to 4 months after treatment. Effective contraception includes surgical sterilization (eg, vasectomy, tubal ligation), two forms of barrier methods (eg, condom, diaphragm) used with spermicide, IUDs, and abstinence.

Exclusion Criteria:

1. Serious uncontrolled concomitant disease that would contraindicate the use of the investigational drug used in this study or that would put the subject at high risk for treatment-related complications.
2. Systemic autoimmune disease (eg, lupus erythematosus, rheumatoid arthritis, Addison's disease, autoimmune disease associated with lymphoma).
3. History of organ transplant requiring immunosuppression.
4. History of or active inflammatory bowel disease (eg, Crohn's disease, ulcerative colitis).
5. Inadequate organ function, evidenced by the following laboratory results:

   1. Absolute neutrophil count < 1,000 cells/mm3.
   2. Platelet count < 75,000 cells/mm3.
   3. Total bilirubin greater than the upper limit of normal (ULN; unless the subject has documented Gilbert's syndrome).
   4. Aspartate aminotransferase (AST [SGOT]) or alanine aminotransferase (ALT [SGPT]) > 2.5 × ULN (> 5 × ULN in subjects with liver metastases).
   5. Alkaline phosphatase levels > 2.5 × ULN (> 5 × ULN in subjects with liver metastases, or >10 × ULN in subjects with bone metastases).
   6. Serum creatinine > 2.0 mg/dL or 177 μmol/L.
   7. Serum anion gap > 16 mEq/L or arterial blood with pH < 7.3.
   8. Medically uncorrectable grade 3 anemia (hemoglobin < 8 g/dL).
6. Uncontrolled hypertension (systolic > 160 mm Hg and/or diastolic > 110 mm Hg) or clinically significant (ie, active) cardiovascular disease, cerebrovascular accident/stroke, or myocardial infarction within 6 months prior to first study medication; unstable angina; congestive heart failure of New York Heart Association grade 2 or higher; or serious cardiac arrhythmia requiring medication. Subjects with uncontrolled hypertension should be medically managed on a stable regimen to control hypertension prior to study entry.
7. Serious myocardial dysfunction defined by ECHO as absolute left ventricular ejection fraction (LVEF) 10% below the institution's lower limit of predicted normal.
8. Dyspnea at rest due to complications of advanced malignancy or other disease requiring continuous oxygen therapy.
9. Positive results of screening test for human immunodeficiency virus (HIV).
10. Current chronic daily treatment (continuous for > 3 months) with systemic corticosteroids (dose equivalent to or greater than 10 mg/day methylprednisolone), excluding inhaled steroids. Short-term steroid use to prevent IV contrast allergic reaction or anaphylaxis in subjects who have known contrast allergies is allowed.
11. Known hypersensitivity to any component of the study medication(s).
12. Subjects taking any medication(s) (herbal or prescribed) known to have an adverse drug reaction with any of the study medications.
13. Concurrent or prior use of a strong cytochrome P450 (CYP)3A4 inhibitor (including ketoconazole, itraconazole, posaconazole, clarithromycin, indinavir, nefazodone, nelfinavir, ritonavir, saquinavir, telithromycin, voriconazole, and grapefruit products) or strong CYP3A4 inducers (including phenytoin, carbamazepine, rifampin, rifabutin, rifapentin, phenobarbital, and St John's Wort) within 14 days before study day 1.
14. Concurrent or prior use of a strong CYP2C8 inhibitor (gemfibrozil) or moderate CYP2C8 inducer (rifampin) within 14 days before study day 1.
15. Participation in an investigational drug study or history of receiving any investigational treatment within 14 days prior to initiation of treatment on this study, except for receipt of testosterone-lowering therapy in men with prostate cancer, or treatment with any NANT Cancer Vaccine therapy.
16. Assessed by the Investigator to be unable or unwilling to comply with the requirements of the protocol.
17. Concurrent participation in any interventional clinical trial.
18. Pregnant and nursing women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2018-07-17 (Actual); Primary Completion 2019-04-17 (Actual); Study Completion 2019-08-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Chan Soon-Shiong Institute for Medicine, El Segundo, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Only the Phase 1b portion of the study enrolled participants. The study was terminated early, so no participants were enrolled on the Phase 2 portion of the study.
  Eligible participants could have gone through both induction and maintenance treatment on study.
Period: Overall Study
Arm/Group | NANT Pancreatic Cancer Vaccine
Started | 3
Completed | 0
Not Completed | 3
Not completed — Progressive Disease | 3

BASELINE CHARACTERISTICS:
Groups:
- NANT Pancreatic Cancer Vaccine: A combination of agents will be administered to subjects in this study: Aldoxorubicin HCl, ALT-803, ETBX-011 (CEA), ETBX-021 (HER2), ETBX-051 (Brachyury), ETBX-061 (MUC1), GI-4000, GI-6207, GI-6301, haNK for infusion, avelumab, bevacizumab, capecitabine, cyclophosphamide, fluorouracil, leucovorin, nab-paclitaxel, oxaliplatin, and Stereotactic Body Radiation Therapy (SBRT).
Arm/Group | NANT Pancreatic Cancer Vaccine
Number analyzed (Participants) | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.3 (5.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
subjects with pancreatic cancer who have progressed on or after standard-of-care therapy [Count of Participants; unit: Participants] | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (AEs) and Serious AEs (SAEs)
Description: Graded Using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03
Time Frame: Up to 230 days
Measure: Count of Participants; unit: Participants
Arm/Group | NANT Pancreatic Cancer Vaccine
Number analyzed (Participants) | 3
Participants
  Treatment-Emergent Adverse Events | 3
  Treatment-Emergent Serious Adverse Events | 2

2. Secondary Outcome: Objective Response Rate by RECIST Version 1.1
Description: Tumors were assessed at screening, and tumor response will be assessed every 8 weeks during the induction phase, and every 12 weeks during the maintenance phase by computed tomography (CT) or magnetic resonance imaging (MRI) of target and non-target lesions in accordance with RECIST Version 1.1.
  An objective response is defined as a confirmed complete or partial overall response with confirmation occurring at least 4 weeks after the initial response is observed.
Time Frame: Tumors were assessed at screening, and tumor response will be assessed every 8 weeks during the induction phase, and every 12 weeks during the maintenance phase until disease progression, up to 6.8 months
Measure: Count of Participants; unit: Participants
Groups:
- NANT Pancreatic Cancer Vaccine: A combination of agents were administered to subjects in this study:
  Aldoxorubicin Hydrochloride
  ALT-803: Recombinant human super agonist interleukin-15 (IL-15) complex
  ETBX-011: Ad5 [E1-, E2b-]-CEA
  ETBX-021: Ad5 [E1-, E2b-]-HER2
  ETBX-051: Ad5 [E1-, E2b-]-Brachyury
  ETBX-061: Ad5 [E1-, E2b-]-MUC1
  GI-4000: RAS yeast
  GI-6207: Carcinoembryonic Antigen (CEA) yeast
  GI-6301: Brachyury yeast
  haNK for infusion: NK-92 [CD16.158V, ER IL-2]
  bevacizumab: Recombinant human anti-Vascular Endothelial Growth Factor (VEGF) IgG1 monoclonal
  Capecitabine: 5'-deoxy-5-fluoro-N-[(pentyloxy) carbonyl]-cytidine
  Cyclophosphamide: 2-[bis(2-chloroethyl)amino]tetrahydro-2H-1,3,2-oxazaphosphorine 2-oxide monohydrate
  Fluorouracil: 5-fluoro-2,4 (1H,3H)-pyrimidinedione
  Leucovorin: L-Glutamic acid, N-[4-[[(2-amino-5-formyl-1,4,5,6,7,8-hexahydro-4-oxo-6-pteridinyl)methyl]amino]benzoyl]-, calcium salt
  nab-Paclitaxel: Benzenepropanoic acid, β-(benzoylamino)-α-hydroxy-(2aR, 4S, 4aS, 6R, 9S, 11S, 12S, 12aR, 12bS)-6,12b-bis(acetyloxy)-12-(benzoyloxy)-2a, 3, 4, 4a, 5, 6, 9, 10, 11, 12, 12a, 12b-dodecahydro-4,11-dihydroxy-4a, 8, 13, 13-tetramethyl-5-oxo-7,11-methano-1H-cyclodeca[3,4]benz[1,2-b]oxet-9-y1ester,(αR,βS)-(9CI) bound to albumin
  Oxaliplatin: cis-[(1 R,2 R)-1,2-cyclohexanediamine-N,N'] [oxalato(2-)- O,O'] platinum
  Avelumab: Recombinant human anti-programmed death-ligand 1 (PD-L1) IgG1 monoclonal antibody
  SBRT: Stereotactic Body Radiation Therapy
Arm/Group | NANT Pancreatic Cancer Vaccine
Number analyzed (Participants) | 3
Participants | 0

3. Secondary Outcome: Objective Response Rate by irRC
Description: Tumors were assessed at screening, and tumor response will be assessed every 8 weeks during the induction phase, and every 12 weeks during the maintenance phase by computed tomography (CT) or magnetic resonance imaging (MRI) of target and non-target lesions in accordance with immune-related response criteria (irRC).
  An objective response is defined as a confirmed complete or partial overall response with confirmation occurring at least 4 weeks after the initial response is observed.
Time Frame: Tumors were assessed at screening, and tumor response will be assessed every 8 weeks during the induction phase, and every 12 weeks during the maintenance phase until confirmed disease progression, up to 6.8 months
Population: No participants had either confirmed partial response or complete response on study. Therefore, objective response rate is 0.
Measure: Count of Participants; unit: Participants
Arm/Group | NANT Pancreatic Cancer Vaccine
Number analyzed (Participants) | 3
Participants | 0

4. Secondary Outcome: Progression Free Survival by RECIST Version 1.1.
Description: PFS was evaluated using Kaplan-Meier methods. PFS was defined as the time from the date of first treatment to the date of disease progression or death (any cause) whichever occurs first. Subjects completing study follow-up or initiating a new anticancer therapy prior to documented PD was censored in the PFS analysis at the last known date the subject was progression free prior to completing follow-up or initiating the new therapy.
Time Frame: Tumors were assessed at screening, and tumor response was assessed every 8 weeks during the induction phase, and every 12 weeks during the maintenance phase until disease progression or death (any cause) whichever occurred first, up to 6.8 months.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | NANT Pancreatic Cancer Vaccine
Number analyzed (Participants) | 3
Months | 1.7 [0.5 to NA] — NA = insufficient number of participants with events.

5. Secondary Outcome: Progression Free Survival by irRC
Description: as for outcome 4
Time Frame: Tumors were assessed at screening, and tumor response was assessed every 8 weeks during the induction phase, and every 12 weeks during the maintenance phase until disease progression or death (any cause) whichever occurred first.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | NANT Pancreatic Cancer Vaccine
Number analyzed (Participants) | 3
Months | 1.7 [0.5 to NA] — NA = insufficient number of participants with events

6. Secondary Outcome: Overall Survival
Description: OS was evaluated using Kaplan-Meier methods. OS was defined as the time from the date of first treatment to the date of death (any cause). Participants who were alive at the end of follow-up were censored in the OS analysis at the last known date alive.
Time Frame: Participants were assessed from screening to death.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | NANT Pancreatic Cancer Vaccine
Number analyzed (Participants) | 3
Months | 4.6 [2.5 to NA] — NA = insufficient number of participants with events

7. Secondary Outcome: Duration of Response (DOR) by RECIST Version 1.1 and irRC
Description: DOR was be defined as the time from the date of first response (PR or CR) to the date of disease progression or death (any cause) whichever occurs first. Responding subjects completed study follow-up or initiating a new anticancer therapy prior to documented PD were censored in the DOR analysis at the last known date the subject was progression free prior completing follow-up or initiating the new therapy.
Time Frame: as for outcome 3
Population: There were no participants with confirmed CR or PR. Therefore, no participants were included in the DOR analysis.
Arm/Group | NANT Pancreatic Cancer Vaccine
Number analyzed (Participants) | 0

8. Secondary Outcome: Disease Control Rate (Confirmed Complete Response, Partial Response, or Stable Disease Lasting for at Least 2 Months) by RECIST Version 1.1 and irRC
Description: Disease control is defined as subjects with a confirmed CR, PR, or SD lasting for at least 2 months.
Time Frame: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | NANT Pancreatic Cancer Vaccine
Number analyzed (Participants) | 3
Participants
  Complete Response | 0
  Partial Response | 0
  Stable Disease | 1

9. Secondary Outcome: Quality of Life by Patient Reported Outcomes (PRO)
Description: PROs were assessed using the Functional Assessment of Cancer Therapy-Hepatobiliary (FACT-Hep) questionnaire. The FACT-Hep is compilation of general questions divided into five QOL subscales:
  Physical Well-Being - Scores ranging from 0-28 Social/Family Well-Being - Scores ranging from 0-28 Emotional Well-Being - Scores ranging from 0-24 Functional Well-Being - Scores ranging from 0-28 Additional Concerns - Scores ranging from 0-72
  It uses 5-point Likert-type response categories ranging from 0 = 'not at all' to 4 = 'very much'
  The higher scales and subscales indicate better quality of life. Negatively worded items were reverse scored. If the missing for each subscale was less than 50%, the prorating scores were computed for the subscale.
Time Frame: 30 days after last dose, up 12.7 months
Population: The questionnaire was not completed for every patient at every visit.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | NANT Pancreatic Cancer Vaccine
Number analyzed (Participants) | 3
score on a scale
  Physical Well-Being - Baseline: number analyzed (Participants) | 2
  Physical Well-Being - Baseline | 13.3 [11.7 to 15.0]
  Physical Well-Being - (I) C3D1: number analyzed (Participants) | 2
  Physical Well-Being - (I) C3D1 | 16.5 [14.0 to 19.0]
  Physical Well-Being - (I) C5D1: number analyzed (Participants) | 1
  Physical Well-Being - (I) C5D1 | 9.0 [9.0 to 9.0]
  Physical Well-Being - (I) C7D1: number analyzed (Participants) | 1
  Physical Well-Being - (I) C7D1 | 11.0 [11.0 to 11.0]
  Physical Well-Being - (I) C9D1: number analyzed (Participants) | 1
  Physical Well-Being - (I) C9D1 | 3.0 [3.0 to 3.0]
  Physical Well-Being - (M) C1D1: number analyzed (Participants) | 1
  Physical Well-Being - (M) C1D1 | 12.0 [12.0 to 12.0]
  Physical Well-Being - End of Treatment: number analyzed (Participants) | 1
  Physical Well-Being - End of Treatment | 22.0 [22.0 to 22.0]
  Social/Family Well-Being - Baseline: number analyzed (Participants) | 2
  Social/Family Well-Being - Baseline | 25.5 [23.0 to 28.0]
  Social/Family Well-Being- (I) C3D1: number analyzed (Participants) | 2
  Social/Family Well-Being- (I) C3D1 | 26.0 [24.0 to 28.0]
  Social/Family Well-Being- (I) C5D1: number analyzed (Participants) | 1
  Social/Family Well-Being- (I) C5D1 | 20.0 [20.0 to 20.0]
  Social/Family Well-Being - (I) C7D1: number analyzed (Participants) | 1
  Social/Family Well-Being - (I) C7D1 | 25.0 [25.0 to 25.0]
  Social/Family Well-Being - (I) C9D1: number analyzed (Participants) | 1
  Social/Family Well-Being - (I) C9D1 | 23.0 [23.0 to 23.0]
  Social/Family Well-Being - (M) C1D1: number analyzed (Participants) | 1
  Social/Family Well-Being - (M) C1D1 | 18.0 [18.0 to 18.0]
  Social/Family Well-Being - End of Treatment: number analyzed (Participants) | 1
  Social/Family Well-Being - End of Treatment | 28.0 [28.0 to 28.0]
  Emotional Well-Being - Baseline: number analyzed (Participants) | 2
  Emotional Well-Being - Baseline | 19.0 [16.0 to 22.0]
  Emotional Well-Being - (I) C3D1: number analyzed (Participants) | 2
  Emotional Well-Being - (I) C3D1 | 20.5 [19.0 to 22.0]
  Emotional Well-Being - (I) C5D1: number analyzed (Participants) | 1
  Emotional Well-Being - (I) C5D1 | 18.0 [18.0 to 18.0]
  Emotional Well-Being - (I) C7D1: number analyzed (Participants) | 1
  Emotional Well-Being - (I) C7D1 | 14.0 [14.0 to 14.0]
  Emotional Well-Being - (I) C9D1: number analyzed (Participants) | 1
  Emotional Well-Being - (I) C9D1 | 13.0 [13.0 to 13.0]
  Emotional Well-Being - (M) C1D1: number analyzed (Participants) | 1
  Emotional Well-Being - (M) C1D1 | 8.0 [8.0 to 8.0]
  Emotional Well-Being - End of Treatment: number analyzed (Participants) | 1
  Emotional Well-Being - End of Treatment | 21.0 [21.0 to 21.0]
  Functional Well-Being - Baseline: number analyzed (Participants) | 2
  Functional Well-Being - Baseline | 15.0 [8.0 to 22.0]
  Functional Well-Being - (I) C3D1: number analyzed (Participants) | 2
  Functional Well-Being - (I) C3D1 | 18.0 [15.0 to 21.0]
  Functional Well-Being - (I) C5D1: number analyzed (Participants) | 1
  Functional Well-Being - (I) C5D1 | 17.0 [17.0 to 17.0]
  Functional Well-Being - (I) C7D1: number analyzed (Participants) | 1
  Functional Well-Being - (I) C7D1 | 12.0 [12.0 to 12.0]
  Functional Well-Being - (I) C9D1: number analyzed (Participants) | 1
  Functional Well-Being - (I) C9D1 | 9.0 [9.0 to 9.0]
  Functional Well-Being - (M) C1D1: number analyzed (Participants) | 1
  Functional Well-Being - (M) C1D1 | 10.0 [10.0 to 10.0]
  Functional Well-Being - End of Treatment: number analyzed (Participants) | 1
  Functional Well-Being - End of Treatment | 20.0 [20.0 to 20.0]
  Additional Concerns - Baseline: number analyzed (Participants) | 2
  Additional Concerns - Baseline | 42.4 [36.0 to 49.0]
  Additional Concerns - (I) C3D1: number analyzed (Participants) | 2
  Additional Concerns - (I) C3D1 | 41.3 [36.0 to 46.6]
  Additional Concerns - (I) C5D1: number analyzed (Participants) | 1
  Additional Concerns - (I) C5D1 | 42.0 [42.0 to 42.0]
  Additional Concerns - (I) C7D1: number analyzed (Participants) | 1
  Additional Concerns - (I) C7D1 | 32.0 [32.0 to 32.0]
  Additional Concerns - (I) C9D1: number analyzed (Participants) | 1
  Additional Concerns - (I) C9D1 | 33.0 [33.0 to 33.0]
  Additional Concerns - (M) C1D1: number analyzed (Participants) | 1
  Additional Concerns - (M) C1D1 | 40.0 [40.0 to 40.0]
  Additional Concerns - End of Treatment: number analyzed (Participants) | 1
  Additional Concerns - End of Treatment | 47.0 [47.0 to 47.0]

ADVERSE EVENTS:
Time Frame: Non-serious AEs were followed for 30 days after the subject's last dose of study treatment, up to 230 days. Non-serious grade 3 or 4 AEs were followed until resolution or stabilization, up to 230 days. All SAEs that had not resolved upon discontinuation of the subject's participation in the study were followed until recovered, recovered with sequelae, not recovered (death due to other cause), death (due to the SAE), lost to follow-up, up to 230 days.
Arm/Group | NANT Pancreatic Cancer Vaccine
All-Cause Mortality (participants affected / at risk) | 3/3
Serious Adverse Events (participants affected / at risk) | 2/3
Other Adverse Events (participants affected / at risk) | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NANT Pancreatic Cancer Vaccine (N=3)
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Disease progression (General disorders) | 1
Clostridium difficile infection (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | NANT Pancreatic Cancer Vaccine (N=3)
Fatigue (General disorders) | 3
Disease progression (General disorders) | 2
Pyrexia (General disorders) | 2
Catheter site haemorrhage (General disorders) | 1
Chills (General disorders) | 1
Gait disturbance (General disorders) | 1
Generalised oedema (General disorders) | 1
Injection site erythema (General disorders) | 1
Injection site reaction (General disorders) | 1
Mucosal dryness (General disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 2
Neutropenia (Blood and lymphatic system disorders) | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Impaired gastric emptying (Gastrointestinal disorders) | 1
Mouth ulceration (Gastrointestinal disorders) | 1
Obstruction gastric (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Clostridium difficile infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 1
Nail injury (Injury, poisoning and procedural complications) | 1
Deep vein thrombosis (Vascular disorders) | 2
Electrocardiogram T wave inversion (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Hyponatraemia (Investigations) | 1
Headache (Nervous system disorders) | 1
Depression (Psychiatric disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-01): https://cdn.clinicaltrials.gov/large-docs/69/NCT03586869/Prot_SAP_000.pdf